# Reducing HIV Vulnerability Through a Multilevel Life Skills Intervention for Adolescent Men: The iREACH

Project Principal Investigators:

Jose Bauermeister, PhD, University of Pennsylvania

Rob Stephenson, PhD, University of Michigan

Patrick Sullivan PhD, Emory University

Protocol identification number: 1U01MD011274-01

ClinicalTrials.gov identifier: NCT03155841

IRB Protocol Number: 825686

Date of Document: March 6, 2019

## Consent to Participate in a Research Study

# *iReach Reducing HIV vulnerability through a multilevel life skills intervention*

Title of the Research Study: Reducing HIV vulnerability through a multilevel life skills

intervention for adolescent men **Protocol Number:** 825686

ClinicalTrials.gov identifier: NCT03155841

**Principal Investigators:** 

Dr. José Bauermeister: 215-898-9993 or bjose@nursing.upenn.edu

**Dr. Rob Stephenson**: 734-615-0149 or rbsteph@umich.edu **Dr. Patrick Sullivan**: 404-727-2038 or pssulli@emory.edu

Study Contact: (James Wolfe, 215-573-4299, jameswol@nursing.upenn.edu)

## What is this study about?

You are invited to be a part of a research study testing a WebApp called iREACH. The purpose of the study is to test whether the iREACH app improves the health and well-being of young men who are attracted to men by helping them to set goals and learn skills to help reach those goals.

This form will give you information to think about before you decide if you want to consent (agree) to be in this study. You get to choose if you want to join the study or not. If you decide to join, you can change your mind later on. You can stop being in the study at any time. We are asking you to participate because you reported that you are a man between the ages of 13 and 18 who reports same-sex attractions.

## What does my participation in this study involve?

If you agree to be part of the study, you will be asked to do two main things: First, you will be asked to complete a survey now, and again every three months for either the next year or the next 15 months. Each survey will take about 30-45 minutes to complete. The survey will ask for general information about you (such as race/ethnicity, income, and education level). It will ask about your health habits, general mood, important relationships in your life, and online habits. It will also ask for sensitive information about your health, sexual behaviors, substance use, and your sexual partner history.

The second main thing we ask you to do is to use a WebApp called iREACH, which you can access on a computer, smartphone, or tablet. iREACH provides a directory of resources for young people. It also includes information on life skills, tools for setting goals, a discussion forum, and the ability to talk to a peer mentor about your goals. Everyone who joins the study

will get access to all the features, but not at the same time. Some people will get access after they sign up, and others will get access a year after signing up. This is decided randomly, like flipping a coin.

If you are randomly chosen to get access to the app right away, your participation will last about a year. If you are randomly chosen to get access to the app after a year's time, your participation will last about 15 months.

## What is the potential risk of participating in this study?

Every research study has risks but there are very little risks involved in this study. Some questions that you will be asked might make you feel uncomfortable. You may skip any survey question you do not want to answer. Also, you are free to leave the research study at any time.

You do not need your parents' approval to join this study. Some people may not be out to their parents and/or want their parents to know that they are in this study. We are taking active steps to protect your privacy. If your parent(s) learn that you're in this study, they will not have access to your answers or experiences you share with us. If you want to tell your parent(s) that you are interested in participating and want them to speak with us, or if they find out about your participation, they can reach us at 833-356-0104.

Your safety is important to us. If you are in trouble and need to talk to crisis counselor, you can call the emergency number at the National Runaway Safeline at any time (1-800-786-2929). iReach also has a special page listing resources you can use. It includes resources for mental health, substance use, and HIV/other sexually transmitted infections. Also, if we learn that you or someone else is at risk for being harmed, we may report this to authorities to protect your safety and the safety of others.

## How will you protect my privacy?

The information we collect in this study is considered confidential, which means that it will be kept private except in specific situations. That includes your survey answers, your use of the iReach WebApp, and even that you are part of this project. To protect your information, we will keep your records filed under a number, not your name or email address. Your records will be kept either in a locked cabinet or on secure computer systems for five years and then will be destroyed.

When you get access to the peer mentoring feature of iREACH, you will be able to chat privately with a peer mentor using a program called VSee. You will get to choose between video, audio, and text chat. Sessions will be recorded and used for supervision of the peer mentors. Only sound and text from sessions will be recorded. Recordings will be deleted after they have been typed into text files.

We will only share your information with specific people. For now, your information will only be shared with the research team which includes the Principal Investigators, and their research staff. We may also store and use your information for future research with other researchers; however, we will not share any information that could identify you.

People other than the researchers may need to see your information. This includes groups that make sure the research is done safely and properly. These groups include the University of Pennsylvania, University of Michigan, Emory University, and the National Institutes of Health who make sure the research is done safely and properly.

To help us protect your privacy, we have a Certificate of Confidentiality from the National Institutes of Health. With this Certificate, we cannot be forced to share information that may identify you, even by a court subpoena (order), in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings. We will use the Certificate to resist any demands for information that would identify you, except as explained below. The Certificate cannot be used to resist a demand for information from personnel of the United States Government that is used for auditing or evaluation of federally funded projects.

You should understand that a Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If an insurer, employer, or other person obtains your written consent to receive research information, then we may not use the Certificate to withhold that information. The Certificate of Confidentiality does not govern the voluntary disclosure of information by you that is not included in the survey, nor does it represent an endorsement of the research by the Secretary of Health and Human Services.

There are times when we may break confidentiality. We will break confidentiality if we think that you are being hurt by an adult or neglected by a caregiver, or if we think that you may hurt yourself or someone else. Depending on the situation, we may report that information to a crisis hotline, a healthcare provider, or local law enforcement, or an adult you trust. If you are in trouble and need to talk to crisis counselor, you can call the

#### National Runaway Safeline: 1-800-786-2929

We will ask for your home and email address. This is so that we can send your compensation, make sure you only fill out the survey once, and get Census data about the area in which you live. Your home address will only be used to get Census data about your neighborhood. Your home address will not be attached to any of your responses, and will be stored in a separate file. We will use your email address to send you an electronic gift card when you complete study surveys. If you agree, we will keep your email address for five years. Identifying information will not be linked to any of your answers. Also, it will not be used to contact you after the study is over, unless you give us permission below.

#### Will I directly benefit from participating in this study?

You may not get any direct benefit from being in this research study. It is possible that you may benefit by learning life skills and accessing the resources provided by iReach. The study may also help other people like you in the future.

## What happens if I do not choose to join the research study?

You get to choose to be in the study or not. The choice is up to you. There is no penalty if you choose not to join the research study. You won't lose benefits or advantages that you have now or that would come to you in the future.

## What if I change my mind regarding my participation in this study?

Participating in this research is voluntary. Even if you decide to join the study now, you may change your mind and stop at any time. If you no longer want to be in the research study, you can contact Dr. José Bauermeister at the University of Pennsylvania by email (bjose@nursing.upenn.edu) and let him know that you do not want to participate any longer. If you stop participating in this study, information that you already gave us will be kept and used, unless you specifically ask for it to be destroyed.

The research team can also end your participation at any time. This may be because you are not following study instructions, or because the study has stopped.

## Will I be paid for being in this study?

You can be paid up to \$205 total for this study. You will be paid \$30 for completing the first survey. You will be paid \$25 for each survey completed in months 3, 6, and 9. You will be paid \$30 for the survey at month 12.

If you are randomly chosen to receive access to the iREACH app after a year, you will have the opportunity to earn \$40 by using the app in different ways. You will also be asked to complete a survey at month 15, for which you will be paid \$30.

We will email you the first Amazon gift card after you have completed the first survey and have created an iReach user account. We will then email you another Amazon gift card after you complete each additional survey. You must complete a survey to receive the gift card, but you can skip any questions you don't want to answer.

If you are offered the opportunity to earn \$40 for using app features and complete the challenge, that gift card will be paid after you complete the study.

#### What will the researchers do with the data?

We plan to publish the results of this study, but will not include any information that could identify you. Your e-mail address, web-survey account, and any other personal identifiers will be stored in a password-protected encrypted server. This information will be destroyed five years after the study is completed. Your survey answers will not be tied to this personal information. All your answers will be kept password-protected computers. By consenting to this research, you allow the researchers to keep and analyze de-identified study data indefinitely.

## Who can I contact if I have questions about the study?

If you have questions, concerns, or complaints regarding the study or if you have any questions about your rights as a research subject, you should speak with the Principal Investigators listed below.

**Dr. José Bauermeister:** 215-898-9993 or bjose@nursing.upenn.edu

**Dr. Rob Stephenson**: 734-615-0149 or rbsteph@umich.edu **Dr. Patrick Sullivan**: 404-727-2038 or pssulli@emory.edu

If you can't reach a member of the research team or want to talk to someone who is not working with the study, you can contact the Office of Regulatory Affairs at the University of Pennsylvania by calling (215) 898-2614.

## **Consent**

Please click the link below to download and read the consent form.

If you agree to the information that we just went over and want to join the study please click the box next to "I agree" and then click the "Next" button to begin the survey.

Thank you so much for your interest and we hope to work with you soon!